CLINICAL TRIAL: NCT03914612
Title: A Phase III Randomized, Placebo-Controlled Study of Pembrolizumab (MK-3475, NSC #776864) in Addition to Paclitaxel and Carboplatin for Measurable Stage III or IVA, Stage IVB or Recurrent Endometrial Cancer
Brief Title: Testing the Addition of the Immunotherapy Drug Pembrolizumab to the Usual Chemotherapy Treatment (Paclitaxel and Carboplatin) in Stage III-IV or Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCI-2019-02186; NCI-2019-02186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY018 (Other: NRG Oncology); NRG-GY018 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Dedifferentiated Carcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Recurrent Endometrial Adenocarcinoma; Recurrent Endometrial Carcinoma; Recurrent Endometrial Clear Cell Adenocarcinoma; Recurrent Endometrial Dedifferentiated Carcinoma; Recurrent Endometrial Endometrioid Adenocarcinoma; Recurrent Endometrial Mixed Cell Adenocarcinoma; Recurrent Endometrial Serous Adenocarcinoma; Recurrent Endometrial Undifferentiated Carcinoma; Stage III Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8; Stage IV Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8
MeSH Terms: conditions — Endometrial Neoplasms; Carcinosarcoma | interventions — Carboplatin; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On February 6, 2023, all patient treatment assignments were unblinded. Patients randomized to Arm I will not receive additional placebo infusions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (placebo, paclitaxel, carboplatin) (Active Comparator): COMBINATION PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo CT scan throughout the study.
  On February 6, 2023, all patient treatment assignments were unblinded. Patients randomized to Arm 1 will not receive additional placebo infusions.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Paclitaxel; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (pembrolizumab, paclitaxel, carboplatin) (Experimental): COMBINATION PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive pembrolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo CT scan throughout the study.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Paclitaxel; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm II (pembrolizumab, paclitaxel, carboplatin)
Other: Placebo Administration — Given IV
  Arms: Arm I (placebo, paclitaxel, carboplatin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well the combination of pembrolizumab, paclitaxel and carboplatin works compared with paclitaxel and carboplatin alone in treating patients with endometrial cancer that is stage III or IV, or has come back after a period of improvement (recurrent). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Paclitaxel and carboplatin are chemotherapy drugs used as part of the usual treatment approach for this type of cancer. This study aims to assess if adding immunotherapy to these drugs is better or worse than the usual approach for treatment of this cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of pembrolizumab (MK-3475) in combination with paclitaxel and carboplatin in patients with advanced stage (measurable stage III or IVA), stage IVB and recurrent endometrial cancer.

SECONDARY OBJECTIVES:

I. To determine the nature, frequency and degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) for each treatment arm.

II. To evaluate blinded independent central review (BICR) assessed or investigator assessed objective response rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by treatment arm and by mismatch repair (MMR) immunohistochemistry (IHC) status in patients who enter the study with measurable disease.

III. To evaluate BICR assessed or investigator assessed duration of response (DOR) by treatment arm and by MMR IHC status in patients who enter the study with measurable disease.

IV. To evaluate the effect of pembrolizumab (MK-3475) on overall survival (OS) in patients with mismatch repair protein proficient (pMMR) or mismatch repair deficiency (dMMR).

V. To determine whether the addition of pembrolizumab (MK-3475) to standard combination chemotherapy is associated with improved patient reported physical function as measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-physical function scale (short form), quality of life as measured with the Functional Assessment of Cancer Therapy (FACT) - Endometrial Trial Outcome Index (En TOI) and worsened fatigue as measured with the PROMIS-Fatigue scale (short form) in the pMMR patients.

VI. To determine concordance between institutional MMR IHC testing and centralized MMR IHC.

EXPLORATORY OBJECTIVES:

I. To explore the correlation between patient-reported physical function as measured with the PROMIS-physical function scale (short form) and quality of life as measure with the FACT-En TOI.

II. To explore whether the addition of pembrolizumab (MK-3475) to standard combination chemotherapy is associated with self-reported neurotoxicity as measured with the FACT/Gynecologic Oncology Group Neurotoxicity (GOG-Ntx) subscale (short) and the extent to which patients differ on their self-reported bother from side effects of cancer therapy in the pMMR patients.

III. To evaluate the efficacy of pembrolizumab (MK-3475) in combination with paclitaxel and carboplatin in patients with advanced stage (measurable stage III or IVA), stage IVB and recurrent endometrial cancer by Programmed Death Ligand 1 (PD-L1) IHC (positive versus [vs] negative).

IV. To assess the association between PD-L1 IHC (positive vs negative) and mismatch repair status (pMMR and dMMR).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

COMBINATION PHASE: Patients receive placebo intravenously (IV) over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease (SD) or partial response (PR) who still have measurable disease may continue treatment for up to a total 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.

On February 6, 2023, all patient treatment assignments were unblinded. Patients randomized to Arm I will not receive additional placebo infusions.

ARM II:

COMBINATION PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo computed tomography (CT) scan throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Measurable stage III, measurable stage IVA, stage IVB (with or without measurable disease) or recurrent (with or without measurable disease) endometrial cancer.
* Pathology report showing results of institutional MMR IHC testing.
* Histologic confirmation of the original primary tumor is required (submission of pathology report(s) is required). Patients with the following histologic types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, dedifferentiated/undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.).
* Submission of tumor specimens for centralized MMR IHC testing is required after Step 1 and before Step 2 registration.
* In patients with measurable disease, lesions will be defined and monitored by RECIST version (v) 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by CT or magnetic resonance imaging (MRI). Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI.
* Patients may have received

  * NO prior chemotherapy for treatment of endometrial cancer OR
  * Prior adjuvant chemotherapy (e.g., paclitaxel/carboplatin alone or as a component of concurrent chemotherapy and radiation therapy [with or without cisplatin]) provided adjuvant chemotherapy was completed >= 12 months prior to STEP 2 registration.
* Patients may have received prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para aortic radiation therapy, intravaginal brachytherapy, and/or palliative radiation therapy. All radiation therapy must be completed at least 4 weeks prior to STEP 2 registration.
* Patients may have received prior hormonal therapy for treatment of endometrial cancer. All hormonal therapy must be discontinued at least three weeks prior to STEP 2 registration.
* Interval or cytoreductive surgery, after start of treatment on this trial, and prior to documentation of disease progression, is NOT permitted.
* Age >= 18.
* Performance status of 0, 1 or 2.
* Platelets >= 100,000/mcl.
* Absolute neutrophil count (ANC) >= 1,500/mcl.
* Creatinine =< 1.5 x institutional/laboratory upper limit of normal (ULN).
* Total serum bilirubin level =< 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN.
* Thyroid stimulating hormone (TSH) within normal limits. If TSH is not within normal range despite no symptoms of thyroid dysfunction, normal Free T4 level is required.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of Step 2 registration are eligible for this trial.
* For patients of child bearing potential: negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.
* Administration of study drugs (pembrolizumab [MK-3475], paclitaxel, carboplatin) may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Women of childbearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from at least 14 days prior to Step 2 registration (for oral contraceptives), during treatment, and for 120 days after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Patients will be considered of nonreproductive potential if they are either:

  * Postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age, a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient); OR
  * Have a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to Step 2 registration; OR
  * Have a congenital or acquired condition that prevents childbearing.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information.

Exclusion Criteria:

* Patients with prior treatment with anti-PD-1, anti-PD-L1 or anti-CTLA-4 therapeutic antibody or other similar agents.
* Patients who have a history of a severe hypersensitivity reaction to monoclonal antibody or pembrolizumab (MK-3475) and/or its excipients; and/or a severe hypersensitivity reaction to paclitaxel and/or carboplatin.
* Patients who are currently participating and receiving cancer-directed study therapy or have participated in a study of an investigational agent and received cancer-directed study therapy within 4 weeks prior to Step 2 registration.
* Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Step 2 registration.

  * Patients who have received steroids as CT scan contrast premedication may be enrolled.
  * The use of inhaled or topical corticosteroids is allowed.
  * The use of mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
  * The use of physiologic doses of corticosteroids may be approved after consultation with the study chair.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression, and they have been off steroids for at least 4 weeks prior to Step 2 registration and remain clinically stable.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. This includes, but is not limited to, patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome because of the risk of recurrence or exacerbation of disease.
* Patients with vitiligo, endocrine deficiencies including type I diabetes mellitus, thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible.
* Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* Patients who have a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection (except for uncomplicated urinary tract infection), interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; and cirrhosis.

  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Pregnant or lactating patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2026-09-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ramez N Eskander, Principal Investigator — NRG Oncology
Locations (397):
- United States (370):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Community Cancer Institute, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Mercy Regional Cancer Center, Redding, California
  - Mercy Oncology Center, Redding, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Bradenton Cancer Center, Bradenton, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Florida Cancer Specialists - Venice Island, Venice, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - WellStar Health System Inc, Marietta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - WellStar North Fulton Hospital, Roswell, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - WellStar Vinings Health Park, Smyrna, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Valley Medical Group - Wayne Multispecialty Practice, Wayne, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Westchester Medical Center, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (14):
  - The Moncton Hospital, Moncton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Japan (4):
  - Ehime University Hospital, Tōon, Ehime
  - Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Saitama Medical University International Medical Center, Saitama
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico
- South Korea (8):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - Samsung Changwon Hospital, Seoul, Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Yonsei University Health System-Severance Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Eskander RN, Sill MW, Beffa L, Moore RG, Hope JM, Musa FB, Mannel RS, Shahin MS, Cantuaria GH, Girda E, Lokich E, Kavecansky J, Leath CA 3rd, Gien LT, Hinchcliff EM, Lele SB, Landrum LM, Backes F, O'Cearbhaill RE, Baghdadi TA, Hill EK, Thaker PH, John VS, Welch S, Fader AN, Powell MA, Aghajanian C. Pembrolizumab plus chemotherapy in advanced or recurrent endometrial cancer: overall survival and exploratory analyses of the NRG GY018 phase 3 randomized trial. Nat Med. 2025 May;31(5):1539-1546. doi: 10.1038/s41591-025-03566-1. Epub 2025 Mar 5. PMID 40044930
- [Derived] Morton M, Marcu I, Levine M, Cosgrove C, Backes F, O'Malley D, Chambers L. Evaluation of Efficacy and Adverse Events After Second Immunotherapy Exposure in Endometrial and Cervical Carcinoma. Obstet Gynecol. 2023 Aug 1;142(2):360-363. doi: 10.1097/AOG.0000000000005243. Epub 2023 Jul 5. PMID 37411031
- [Derived] Eskander RN, Sill MW, Beffa L, Moore RG, Hope JM, Musa FB, Mannel R, Shahin MS, Cantuaria GH, Girda E, Mathews C, Kavecansky J, Leath CA 3rd, Gien LT, Hinchcliff EM, Lele SB, Landrum LM, Backes F, O'Cearbhaill RE, Al Baghdadi T, Hill EK, Thaker PH, John VS, Welch S, Fader AN, Powell MA, Aghajanian C. Pembrolizumab plus Chemotherapy in Advanced Endometrial Cancer. N Engl J Med. 2023 Jun 8;388(23):2159-2170. doi: 10.1056/NEJMoa2302312. Epub 2023 Mar 27. PMID 36972022

RESULTS

PARTICIPANT FLOW:
Groups:
- (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin); (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin): COMBINATION PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity. MAINTENANCE PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.
- (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin); (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin): COMBINATION PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity. MAINTENANCE PHASE: Patients receive pembrolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Started | 113 | 112 | 295 | 293
Completed | 113 | 112 | 295 | 293
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population (with definitive MMR status)
Groups:
- Total: Total of all reporting groups
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | Total
Number analyzed (Participants) | 113 | 112 | 295 | 293 | 813
Age, Continuous [Median (Full Range); unit: years] | 66 [37 to 85] | 67 [38 to 81] | 65 [29 to 90] | 66 [31 to 93] | 66 [29 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 112 | 295 | 293 | 813
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 16 | 21 | 48
  Not Hispanic or Latino | 99 | 106 | 273 | 263 | 741
  Unknown or Not Reported | 8 | 1 | 6 | 9 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 2 | 6
  Asian | 4 | 3 | 14 | 17 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 3 | 1 | 4
  Black or African American | 9 | 11 | 51 | 45 | 116
  White | 86 | 92 | 212 | 212 | 602
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 12 | 6 | 12 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) Note: For arm 2 (dMMR Cohort), the point estimate and the upper limit of the confidence interval are not able to be estimated due to insufficient events.
Time Frame: Duration of time from study entry to time of progression per RECIST criteria or death due to any cause, whichever occurs first. The interquartile range for follow-up was (6.37 months, 30.62 months). The maximum for follow-up was 37.85 months.
Population: Randomized population (with determinate MMR status)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 113 | 112 | 295 | 293
Months | 7.6 [6.4 to 9.9] | NA [30.6 to NA] — The point estimate and the upper limit of the confidence interval are not able to be estimated due to insufficient events. | 8.7 [8.4 to 10.7] | 11.7 [11.0 to 15.0]

2. Secondary Outcome: Adverse Events With Grade 3 (or Higher)
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE V5.0). The endpoint is the count of participants with an adverse event of grade 3 (or higher) by treatment group.
Time Frame: For the adverse event time frame, the interquartile range was (0.79 months, 3.42 months); the maximum was 28.39 months.
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 106 | 109 | 274 | 276
Participants | 50 | 68 | 124 | 151

3. Secondary Outcome: Objective Tumor Response
Description: Assessed by Response Evaluation Criteria for Solid Tumors (RECIST) 1.1.
Time Frame: For the time frame for tumor response, the interquartile range was (2.27 months, 8.66 months) and the maximum was 36.37 months.
Population: Randomized patients with measurable disease
Measure: Count of Participants; unit: Participants
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 92 | 92 | 234 | 212
Participants | 65 | 75 | 136 | 150

4. Secondary Outcome: Duration of Objective Response
Description: The time difference between the dates of first response and first progression; patients who do not progress are considered censored. Note: for Arm 2 (dMMR Cohort), the upper limit of the confidence interval is not able to be estimated due to an insufficient number of events.
Time Frame: For the duration of objective response, the interquartile range is (4.24 months, 7.92 months); the maximum is 28.68 months.
Population: Randomized patients with objective tumor response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 65 | 75 | 136 | 150
Months | 6.2 [4.3 to 9.2] | 28.7 [20.2 to NA] — The upper limit of the confidence interval is not able to be estimated due to an insufficient number of events. | 6.2 [4.8 to 6.5] | 9.2 [7.1 to 14.7]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS). This endpoint will be assessed by Kaplan-Meier.
Time Frame: Time from study entry to time of death or the date of last contact, assessed up to 5 years
Reporting Status: Not Posted, anticipated posting 2029-04

6. Secondary Outcome: Quality of Life (QoL) in pMMR Patients Only
Description: QoL are collected in pMMR patients only and measured with the Function Assessment of Cancer Therapy -Endometrial Trial Outcome Index (FACT En-TOI). The FACT-En TOI scores range 0 - 120 with a larger score suggesting better or favorable state of QOL.
Time Frame: 0-54 weeks from start of treatment
Population: The pMMR patients who provided baseline and at least one follow-up QOL assessment.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 254 | 248
score
  Baseline | 94.5 (18.0) | 95.3 (16.7)
  6 weeks: number analyzed (Participants) | 249 | 239
  6 weeks | 94.1 (15.1) | 92.0 (15.5)
  18 weeks: number analyzed (Participants) | 212 | 218
  18 weeks | 93.4 (15.5) | 90.3 (16.2)
  30 weeks: number analyzed (Participants) | 183 | 196
  30 weeks | 95.7 (16.6) | 94.6 (15.7)
  54 weeks: number analyzed (Participants) | 142 | 149
  54 weeks | 93.5 (18.2) | 96.8 (15.0)

7. Secondary Outcome: Concordance Between Institutional Mismatch Repair (MMR) Immunohistochemistry (IHC) Testing and Centralized MMR IHC
Description: Concordance between institutional MMR IHC testing and centralized MMR IHC. The concordance of institutional MMR IHC testing and centralized MMR IHC will be characterized by agreement statistics including the kappa statistic (e.g. Cohen's kappa coefficient).
Time Frame: IHC testing values (for both central and institutional) were collected at baseline.
Population: Patients from Japan were excluded. Otherwise all patients with a valid institutional MMR IHC status and a valid centralized MMR IHC status at baseline.
Measure: Number (95% Confidence Interval); unit: agreement score
Groups:
- Arm I: Active Comparator (Placebo, Paclitaxel, Carboplatin): COMBINATION PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity. MAINTENANCE PHASE: Patients receive placebo IV over 30 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.
- Arm II: Experimental (Pembrolizumab, Paclitaxel, Carboplatin): COMBINATION PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle, paclitaxel IV over 3 hours on day 1 of each cycle, and carboplatin IV over 30 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease may continue treatment for up to a total of 10 cycles (if deemed necessary by the treating physician) in the absence of disease progression or unacceptable toxicity. MAINTENANCE PHASE: Patients receive pembrolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 6 weeks for up to 14 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I: Active Comparator (Placebo, Paclitaxel, Carboplatin) | Arm II: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 375 | 377
agreement score | 0.9197 [0.875 to 0.9644] | 0.8944 [0.8438 to 0.945]

8. Other Pre Specified Outcome: Incidence of Pembrolizumab Treatment and Self-reported Neurotoxicity
Description: Patient-reported neurotoxicity will be measured with FACT/GOG-Ntx subscale (short form).
Time Frame: 0-54 weeks from start of treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Effect of Pembrolizumab on PFS and OS by Program Death Ligand 1 (PD-L1) IHC
Description: Will assess the effect of pembrolizumab on PFS and OS by PD-L1 (combined positive score [CPS]) within proficient MMR (pMMR) and deficient MMR (dMMR) populations. The effectiveness of pembrolizumab will be compared by PD-L1 status (CPS). A formal test will be conducted by examining the interaction term between pembrolizumab treatment (yes or no) with PD-L1 status. The association between PD-L1 CPS status and MMR IHC status will be assessed with odds ratios. A test may be conducted with a Fisher's Exact Test, and confidence intervals will be provided.
Time Frame: 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Association Between PD-L1 IHC and MMR Status
Description: Measures of association between PD-L1 IHC (CPS) and MMR IHC status. The concordance of institutional MMR IHC testing and centralized MMR IHC will be characterized by agreement statistics such as kappa statistics (e.g. Cohen's kappa coefficient).
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 28.39 months; the interquartile range was (0.79 months, 3.42 months). All-Cause Mortality monitored/assessed up to 37.85 months; the interquartile range was (6.37 months, 30.62 months).
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE). All Enrolled participants monitored/assessed for All-Cause Mortality; participants that received intervention (safety population) monitored/assessed for Serious and Other (Not Including Serious) Adverse Events.
Arm/Group | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 16/113 | 7/112 | 47/295 | 42/293
Serious Adverse Events (participants affected / at risk) | 50/106 | 66/109 | 125/274 | 152/276
Other Adverse Events (participants affected / at risk) | 105/106 | 107/109 | 256/274 | 258/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) (N=106) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) (N=109) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) (N=274) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) (N=276)
Anemia (Blood and lymphatic system disorders) | 10 | 20 | 25 | 38
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 4 | 9
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1 | 1 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0 | 2
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 1
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial tamponade (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 5 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 3 | 4
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 3
Rectal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 3
Fatigue (General disorders) | 4 | 1 | 7 | 5
Fever (General disorders) | 2 | 1 | 2 | 5
Gait disturbance (General disorders) | 0 | 1 | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 | 0 | 0
Generalized edema (General disorders) | 0 | 0 | 0 | 2
Localized edema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 4 | 2
Sudden death NOS (General disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 1 | 1
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 3
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 1 | 4
Kidney infection (Infections and infestations) | 1 | 1 | 1 | 0
Lung infection (Infections and infestations) | 1 | 4 | 0 | 4
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 1 | 3 | 7
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 5 | 9 | 10
Uterine infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 4 | 4 | 4
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 1 | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 2 | 4
INR increased (Investigations) | 0 | 0 | 0 | 2
Investigations - Other, specify (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 8 | 6 | 8 | 16
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 18 | 13 | 32 | 50
Platelet count decreased (Investigations) | 2 | 5 | 6 | 12
Weight gain (Investigations) | 1 | 1 | 0 | 1
Weight loss (Investigations) | 1 | 1 | 2 | 1
White blood cell decreased (Investigations) | 12 | 8 | 17 | 25
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 3 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 8 | 9 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 1 | 2
Myasthenia gravis (Nervous system disorders) | 0 | 2 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 5 | 5 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 2
Seizure (Nervous system disorders) | 0 | 2 | 1 | 4
Stroke (Nervous system disorders) | 1 | 2 | 0 | 0
Syncope (Nervous system disorders) | 6 | 6 | 8 | 7
Transient ischemic attacks (Nervous system disorders) | 0 | 1 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1 | 4
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 1 | 4
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 2 | 0 | 2
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 4 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 0 | 1
Arterial thromboembolism (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 6 | 9 | 13 | 13
Hypotension (Vascular disorders) | 1 | 2 | 1 | 3
Thromboembolic event (Vascular disorders) | 2 | 7 | 12 | 11
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (dMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) (N=106) | (dMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) (N=109) | (pMMR Cohort): Arm 1: Active Comparator (Placebo, Paclitaxel, Carboplatin) (N=274) | (pMMR Cohort): Arm 2: Experimental (Pembrolizumab, Paclitaxel, Carboplatin) (N=276)
Anemia (Blood and lymphatic system disorders) | 58 | 63 | 144 | 152
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 2 | 7 | 5
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 4 | 9
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 4 | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 1 | 1 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 2 | 2 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 2 | 0 | 5
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 1
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 4 | 2 | 6
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1
Pericardial tamponade (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 8 | 13 | 16
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 4 | 4
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 3
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 2 | 6 | 11
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 1 | 2
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 4
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 3 | 3
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 1 | 10 | 10 | 16
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 10 | 14 | 7 | 37
Blurred vision (Eye disorders) | 8 | 11 | 16 | 28
Cataract (Eye disorders) | 0 | 1 | 0 | 2
Dry eye (Eye disorders) | 2 | 5 | 5 | 10
Eye disorders - Other, specify (Eye disorders) | 3 | 5 | 5 | 5
Eye pain (Eye disorders) | 2 | 2 | 2 | 1
Eyelid function disorder (Eye disorders) | 0 | 1 | 0 | 0
Flashing lights (Eye disorders) | 0 | 1 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 1
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Papilledema (Eye disorders) | 0 | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 2 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 1 | 1
Vision decreased (Eye disorders) | 0 | 0 | 0 | 1
Watering eyes (Eye disorders) | 2 | 0 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 7 | 6
Abdominal pain (Gastrointestinal disorders) | 14 | 19 | 45 | 48
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Belching (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 3 | 3 | 8 | 6
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 7 | 4 | 4
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 40 | 47 | 106 | 120
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 36 | 46 | 88 | 99
Dry mouth (Gastrointestinal disorders) | 1 | 11 | 7 | 12
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 5 | 12 | 16
Dysphagia (Gastrointestinal disorders) | 4 | 4 | 2 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Flatulence (Gastrointestinal disorders) | 2 | 3 | 0 | 4
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 3 | 6 | 11
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 | 7 | 7 | 11
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 5
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 4 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 15 | 19 | 12 | 26
Nausea (Gastrointestinal disorders) | 44 | 55 | 114 | 121
Oral cavity fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 5
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2 | 4 | 7
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Stomach pain (Gastrointestinal disorders) | 1 | 3 | 3 | 5
Toothache (Gastrointestinal disorders) | 0 | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 9 | 22 | 38 | 53
Chills (General disorders) | 2 | 7 | 4 | 10
Edema face (General disorders) | 0 | 0 | 1 | 2
Edema limbs (General disorders) | 13 | 13 | 25 | 43
Edema trunk (General disorders) | 0 | 0 | 2 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 59 | 78 | 165 | 175
Fever (General disorders) | 5 | 11 | 8 | 16
Flu like symptoms (General disorders) | 4 | 0 | 1 | 6
Gait disturbance (General disorders) | 3 | 4 | 3 | 7
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 7 | 4 | 6
Generalized edema (General disorders) | 0 | 1 | 1 | 3
Hypothermia (General disorders) | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 2
Localized edema (General disorders) | 2 | 4 | 4 | 5
Malaise (General disorders) | 2 | 0 | 4 | 4
Neck edema (General disorders) | 2 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 5 | 9 | 10
Pain (General disorders) | 11 | 14 | 25 | 39
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 3 | 5 | 12 | 3
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 3
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 1
Immune system disorders - Other, specify (Immune system disorders) | 0 | 0 | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 1
Bladder infection (Infections and infestations) | 1 | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 3
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 1 | 2
Esophageal infection (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 2 | 4 | 6 | 8
Herpes simplex reactivation (Infections and infestations) | 0 | 3 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 12 | 8 | 19 | 23
Kidney infection (Infections and infestations) | 1 | 1 | 2 | 0
Lip infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 4 | 0 | 6
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 1 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 2
Papulopustular rash (Infections and infestations) | 0 | 2 | 2 | 5
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 1 | 1
Sepsis (Infections and infestations) | 3 | 2 | 3 | 7
Shingles (Infections and infestations) | 0 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 3 | 3 | 8
Skin infection (Infections and infestations) | 4 | 4 | 7 | 8
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Thrush (Infections and infestations) | 0 | 1 | 4 | 4
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 3
Upper respiratory infection (Infections and infestations) | 3 | 6 | 4 | 7
Urinary tract infection (Infections and infestations) | 9 | 15 | 32 | 38
Uterine infection (Infections and infestations) | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 2 | 9 | 5
Vulval infection (Infections and infestations) | 0 | 1 | 1 | 1
Wound infection (Infections and infestations) | 1 | 1 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 3 | 8 | 9 | 7
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 10 | 16 | 22
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 6
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 16 | 16 | 35 | 41
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 14 | 16 | 27 | 40
Alkaline phosphatase increased (Investigations) | 17 | 15 | 33 | 35
Aspartate aminotransferase increased (Investigations) | 6 | 13 | 20 | 38
Blood bicarbonate decreased (Investigations) | 0 | 2 | 1 | 2
Blood bilirubin increased (Investigations) | 2 | 6 | 6 | 8
Blood corticotrophin decreased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 2 | 2 | 1 | 2
Cardiac troponin T increased (Investigations) | 0 | 0 | 0 | 2
Cholesterol high (Investigations) | 0 | 1 | 1 | 3
Creatinine increased (Investigations) | 8 | 24 | 24 | 45
GGT increased (Investigations) | 0 | 0 | 1 | 2
Hemoglobin increased (Investigations) | 0 | 2 | 1 | 0
INR increased (Investigations) | 2 | 0 | 2 | 3
Investigations - Other, specify (Investigations) | 1 | 5 | 8 | 10
Lipase increased (Investigations) | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 24 | 24 | 48 | 58
Lymphocyte count increased (Investigations) | 1 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 34 | 28 | 72 | 87
Platelet count decreased (Investigations) | 31 | 38 | 58 | 83
Serum amylase increased (Investigations) | 0 | 0 | 0 | 4
Thyroid stimulating hormone increased (Investigations) | 2 | 3 | 8 | 13
Weight gain (Investigations) | 4 | 7 | 7 | 9
Weight loss (Investigations) | 6 | 16 | 21 | 19
White blood cell decreased (Investigations) | 38 | 35 | 79 | 78
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 19 | 29 | 60 | 54
Dehydration (Metabolism and nutrition disorders) | 8 | 10 | 15 | 12
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 4 | 10 | 14
Hyperglycemia (Metabolism and nutrition disorders) | 23 | 26 | 61 | 61
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 1 | 14 | 10
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 4
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 17 | 27 | 38
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 11 | 19 | 17
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 3 | 8 | 3
Hypokalemia (Metabolism and nutrition disorders) | 21 | 21 | 47 | 37
Hypomagnesemia (Metabolism and nutrition disorders) | 15 | 23 | 50 | 53
Hyponatremia (Metabolism and nutrition disorders) | 8 | 19 | 31 | 37
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 | 1 | 4 | 9
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 32 | 75 | 62
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 15 | 30 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 14 | 27 | 24
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Chest wall necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 8 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 | 14 | 20 | 29
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 7 | 7 | 8 | 11
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 7
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 29 | 46 | 45
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 7 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 12 | 34 | 38
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 1 | 1 | 2
Anosmia (Nervous system disorders) | 1 | 0 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 3
Brachial plexopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 2 | 0 | 0 | 2
Concentration impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 17 | 23 | 35 | 40
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Dysesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 16 | 14 | 33 | 34
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 2 | 4 | 5 | 3
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 18 | 21 | 29 | 42
Lethargy (Nervous system disorders) | 0 | 1 | 2 | 0
Memory impairment (Nervous system disorders) | 4 | 1 | 8 | 4
Movements involuntary (Nervous system disorders) | 0 | 0 | 0 | 2
Muscle weakness left-sided (Nervous system disorders) | 0 | 2 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 1 | 2
Myasthenia gravis (Nervous system disorders) | 0 | 2 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 3 | 6 | 2 | 9
Neuralgia (Nervous system disorders) | 1 | 4 | 3 | 3
Paresthesia (Nervous system disorders) | 7 | 10 | 18 | 16
Peripheral motor neuropathy (Nervous system disorders) | 8 | 12 | 16 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 66 | 71 | 157 | 153
Presyncope (Nervous system disorders) | 1 | 4 | 6 | 3
Seizure (Nervous system disorders) | 0 | 2 | 1 | 4
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Spasticity (Nervous system disorders) | 0 | 0 | 1 | 0
Stroke (Nervous system disorders) | 1 | 2 | 1 | 1
Syncope (Nervous system disorders) | 6 | 6 | 8 | 7
Transient ischemic attacks (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 3 | 4 | 5
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 11 | 16 | 26 | 28
Confusion (Psychiatric disorders) | 1 | 3 | 5 | 7
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 6 | 5 | 7 | 7
Hallucinations (Psychiatric disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 10 | 17 | 29 | 30
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 1 | 8
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 1 | 5
Bladder spasm (Renal and urinary disorders) | 0 | 2 | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 2 | 1 | 6
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 5 | 10 | 13
Glucosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 1 | 6 | 10
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1 | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 6 | 4 | 5
Renal calculi (Renal and urinary disorders) | 0 | 0 | 2 | 1
Urinary frequency (Renal and urinary disorders) | 3 | 6 | 7 | 15
Urinary incontinence (Renal and urinary disorders) | 5 | 11 | 11 | 11
Urinary retention (Renal and urinary disorders) | 0 | 1 | 4 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 4 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 2 | 3
Urinary urgency (Renal and urinary disorders) | 1 | 4 | 7 | 11
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 2 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 2 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 1 | 8 | 7
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 1 | 3 | 3
Uterine fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 3 | 5 | 8 | 7
Vaginal dryness (Reproductive system and breast disorders) | 1 | 1 | 1 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 7 | 4 | 8 | 10
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 2
Vaginal perforation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 6 | 11
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 19 | 38 | 38
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 30 | 52 | 57
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 9 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 6
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 6 | 3
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 9 | 6
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 63 | 62 | 143 | 136
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 8 | 9 | 19
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2
Hair color changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 5 | 4 | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 7
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 6
Nail loss (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 17 | 23 | 39
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 10 | 16 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 34 | 27 | 57
Scalp pain (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 | 7 | 23 | 25
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 9
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 5
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1 | 1 | 4
Arterial thromboembolism (Vascular disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 6 | 10 | 9
Hematoma (Vascular disorders) | 1 | 2 | 0 | 3
Hot flashes (Vascular disorders) | 7 | 8 | 9 | 12
Hypertension (Vascular disorders) | 17 | 23 | 45 | 34
Hypotension (Vascular disorders) | 5 | 5 | 8 | 7
Lymphedema (Vascular disorders) | 0 | 1 | 4 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 3 | 0
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 3 | 12 | 23 | 23
Vascular disorders - Other, specify (Vascular disorders) | 2 | 1 | 3 | 4
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT03914612/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03914612/ICF_001.pdf